CLINICAL TRIAL: NCT02724761
Title: Prophylactic Racemic Epinephrine for the Prevention of Dysphagia in Patients Undergoing Anterior Cervical Discectomy and Fusion: A Randomized Control Trial
Brief Title: Prophylactic Racemic Epinephrine in Anterior Cervical Discectomy and Fusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Andrew Chung (Other)
Collaborators: More Foundation (Other); Banner Health (Other)
Responsible Party: Sponsor-Investigator, Andrew Chung, Co-Investigator, Resident Physician, Banner Health
Organization: Banner Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BannerHealth
Record Dates: First submitted 2016-03-07; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Dysphagia; Dysphonia; Postoperative Pain
MeSH Terms: conditions — Deglutition Disorders; Dysphonia; Pain, Postoperative | interventions — Racepinephrine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Racemic Epinephrine (Experimental): Over the Counter (OTC) - 0.5 mL Nebulized Racemic Epinephrine
  Interventions: Drug: Racemic Epinephrine
- Placebo: 0.9% Normal Saline (Placebo Comparator): 0.5 mL 0.9% Normal Saline
  Interventions: Drug: Placebo (for racemic epinephrine)

INTERVENTIONS:
Drug: Racemic Epinephrine — 1 inhalation of 0.5 mL of 2.25% Nebulized Racemic Epinephrine every 8 hours for 24 hours after surgery
  Other Names: AsthmaNefrin
  Arms: Experimental: Racemic Epinephrine
Drug: Placebo (for racemic epinephrine) — 0.5 mL of normal saline will be prepared in an identical amber syringe as the drug intervention (racemic epinephrine)
  Other Names: 0.9% normal saline
  Arms: Placebo: 0.9% Normal Saline

SUMMARY:
Our double-blinded, randomized control trial will assess the effect of nebulized racemic epinephrine inpatients undergoing anterior cervical discectomy and fusion (ACDF) procedures. The investigators have had success in managing post-operative dysphagia in patients undergoing ACDF with the administration of this drug. Half of the participants will review nebulized epinephrine. The other half will receive placebo.

DETAILED DESCRIPTION:
Based on data from the National Inpatient Sample from 2002-2012, patients undergoing elective primary ACDF, diagnosed with dysphagia (4% of total patients), had a two-fold increase in mean length of stay (4.03 compared to 1.56 days; p < 0.001) and a substantial increase in their total hospital charges (p < 0.001) versus those not diagnosed with dysphagia. There are very few level I studies which describe successful management of these complications. Steroids have shown promise, however, there exist concerns for consequent delayed bony fusion. Racemic epinephrine is a mixture of both the R and L isomers of epinephrine which theoretically results in a milder side effect profile and longer shelf-life versus the standard L-epinephrine. Traditionally, racemic epinephrine has been administered in a nebulized form for the treatment of severe asthma, laryngeal edema, and bronchiolitis. The most severe side effects that have been reported include tachyarrhythmias and paradoxical bronchospasms, although these reports are rare and limited mainly to single case reports or case series. It confers its therapeutic effect through Racemic α-adrenergic and β-adrenergic mediated vasoconstriction of mucosal vasculature decreasing edema and in the respiratory tract, inducing bronchodilation. The PI, has been utilizing nebulized racemic epinephrine at standard dosages (1 unit of 0.5 ml of 2.25% racemic epinephrine) for the treatment of severe post-operative dysphagia in patients undergoing ACDF for 20 years. The investigator has achieved marked success with this intervention with no notable associated complications. Despite being successfully utilized in this manner for many years in small pockets of the spine community, the use of prophylactic racemic epinephrine for the management of dysphagia has not been described in the literature. The investigators hope to be able to fill this important knowledge-gap with our study data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age
2. Primary two and three-level ACDF between C3-7
3. Approved pre-authorization to undergo the procedure

Exclusion Criteria:

1. Patients < 18 years of age
2. Patients who are unable to give their own consent
3. Revision ACDF
4. Combined anterior-posterior surgeries
5. Surgeries involving C2-C3 or C7-T1
6. Surgeries related to trauma, infection, or tumor
7. Patients with baseline swallowing dysfunction
8. Patients currently on steroids
9. Patients with severe cardiac disease
10. Uncontrolled diabetics as defined by patients with a HbA1C > 8%
11. Patients with known allergy to epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in Dysphagia Numeric Rating Scale (DNRS) | Post-operative day 1, just prior to hospital discharge (up to 1 week post-operatively), the first post-operative visit (10-14 days post-operatively, up to 30 days from surgery depending on clinical course).
  It is a simple questionnaire that is a functional assessment of dysphagia i.e. difficulty swallowing solids, liquids, etc. Additionally, asks a simple "yes" and "no" question for the presence of dysphagia.
Change in Visual Analogue Scale (VAS) - Odynophagia | Post-operative day 1, just prior to hospital discharge (up to 1 week post-operatively), the first post-operative visit (10-14 days post-operatively, up to 30 days from surgery depending on clinical course).
  It is a simple self-reported pain intensity scale from 0-10 with 0 being no pain, and 10 being the worst pain possible as it relates to swallowing.

SECONDARY OUTCOMES:
Change in Rate of dysphonia | Post-operative day 1, just prior to hospital discharge (up to 1 week post-operatively), the first post-operative visit (10-14 days post-operatively, up to 30 days from surgery depending on clinical course).
  Patients will be asked to answer whether or not they are experiencing dysphonia with a simple "yes" or "no".
Airway complication | Up to 1 month post-operatively
  Any airway complication related to post-operative swelling that requires intubation will be retrospectively recorded off of hospital records. This will be recorded as the number of patients requiring intubation. This number will be reported in any future presentation of data.
Length of Stay | Up to 30 days post-operatively.
  Length of hospital stay following surgery
Hospital Cost | Up to 30 days post-operatively.
  Will determine any additional cost of care associated with dysphagia, dysphonia, airway complications. This will include any emergency department visits or hospital re-admissions directly related to these post-operative complications.
30-day Hospital re-admission rates | Up to 30 days post-operatively.
  any re-admission in the first 30 days following surgery specifically due to dysphagia, dysphonia, or airway complications related to surgery.
Number of emergency department visits per patient related to surgical complications of dysphagia or difficulty breathing | 30 days
  Number of emergency department visits in the first 30 days following surgery with patient complaint of "difficulty or pain with swallowing" or "difficulty breathing" as direct complications of surgery (i.e. secondary to post-operative swelling, hematoma formation). Patient charts will be retrospectively reviewed 30 days post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Chutkan, MD, Principal Investigator — The CORE Institute, Banner University Medical Center
Locations (1):
- Banner University Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be be presented in a research paper format and submitted to a journal following completion of the study.

REFERENCES:
- [Background] Kalb S, Reis MT, Cowperthwaite MC, Fox DJ, Lefevre R, Theodore N, Papadopoulos SM, Sonntag VK. Dysphagia after anterior cervical spine surgery: incidence and risk factors. World Neurosurg. 2012 Jan;77(1):183-7. doi: 10.1016/j.wneu.2011.07.004. Epub 2011 Nov 15. PMID 22155226
- [Background] Jeyamohan SB, Kenning TJ, Petronis KA, Feustel PJ, Drazin D, DiRisio DJ. Effect of steroid use in anterior cervical discectomy and fusion: a randomized controlled trial. J Neurosurg Spine. 2015 Aug;23(2):137-43. doi: 10.3171/2014.12.SPINE14477. Epub 2015 May 1. PMID 25932600
- [Background] Bazaz R, Lee MJ, Yoo JU. Incidence of dysphagia after anterior cervical spine surgery: a prospective study. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2453-8. doi: 10.1097/00007632-200211150-00007. PMID 12435974
- [Background] Singh K, Marquez-Lara A, Nandyala SV, Patel AA, Fineberg SJ. Incidence and risk factors for dysphagia after anterior cervical fusion. Spine (Phila Pa 1976). 2013 Oct 1;38(21):1820-5. doi: 10.1097/BRS.0b013e3182a3dbda. PMID 23873236
- [Background] Lee MJ, Bazaz R, Furey CG, Yoo J. Risk factors for dysphagia after anterior cervical spine surgery: a two-year prospective cohort study. Spine J. 2007 Mar-Apr;7(2):141-7. doi: 10.1016/j.spinee.2006.02.024. Epub 2007 Jan 22. PMID 17321961
- [Background] Lee SH, Kim KT, Suk KS, Park KJ, Oh KI. Effect of retropharyngeal steroid on prevertebral soft tissue swelling following anterior cervical discectomy and fusion: a prospective, randomized study. Spine (Phila Pa 1976). 2011 Dec 15;36(26):2286-92. doi: 10.1097/BRS.0b013e318237e5d0. PMID 22020609
- [Background] Song KJ, Lee SK, Ko JH, Yoo MJ, Kim DY, Lee KB. The clinical efficacy of short-term steroid treatment in multilevel anterior cervical arthrodesis. Spine J. 2014 Dec 1;14(12):2954-8. doi: 10.1016/j.spinee.2014.06.005. Epub 2014 Jun 12. PMID 24929058
- [Background] Plint AC, Osmond MH, Klassen TP. The efficacy of nebulized racemic epinephrine in children with acute asthma: a randomized, double-blind trial. Acad Emerg Med. 2000 Oct;7(10):1097-103. doi: 10.1111/j.1553-2712.2000.tb01258.x. PMID 11015240
- [Background] Langley JM, Smith MB, LeBlanc JC, Joudrey H, Ojah CR, Pianosi P. Racemic epinephrine compared to salbutamol in hospitalized young children with bronchiolitis; a randomized controlled clinical trial [ISRCTN46561076]. BMC Pediatr. 2005 May 5;5(1):7. doi: 10.1186/1471-2431-5-7. PMID 15876347